CLINICAL TRIAL: NCT00729742
Title: A Phase 1b, Multicenter Trial to Evaluate Molecular Determinants of Response to Erlotinib and MK0646 in Advanced Non-Small-Cell Lung Cancer
Brief Title: Phase I Imaging Study Evaluating Dalotuzumab (MK0646) in Combination With Erlotinib for Patients With Non-Small Cell Lung Cancer (MK-0646-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0646-008; 2008_518; CTRI/2009/091/000139 (Registry Identifier: CTRI)
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Carcinoma, Non-small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dalotuzumab; Erlotinib Hydrochloride

ARMS (2):
- Part 1 (Experimental): erlotinib
  Interventions: Drug: Comparator: erlotinib monotherapy
- Part 2 (Experimental): erlotinib + dalotuzumab
  Interventions: Drug: Comparator: erlotinib + dalotuzumab

INTERVENTIONS:
Drug: Comparator: erlotinib + dalotuzumab — Part II: All patients will receive 1 week of erlotinib 150 mg tablets per day.
  Arm 1: Patients who experience a PET response will continue on erlotinib monotherapy until disease progression.
  Arm 2: Patients who fail to receive a PET response will continue to take erlotinib in combination with dalotuzumab 10 mg/kg IV infusion once weekly. At the time of disease progression, patients on erlotinib monotherapy will be offered to crossover to dalotuzumab 10 mg/kg IV infusion once weekly in combination with erlotinib.
  Other Names: TARCEVA®
  Arms: Part 2
Drug: Comparator: erlotinib monotherapy — Part I: All patients will receive erlotinib 150 mg tablets per day until disease progression.
  Other Names: TARCEVA®
  Arms: Part 1

SUMMARY:
This study will use imaging to look at tumor response to erlotinib (Part I) and the combination of erlotinib and dalotuzumab (Part II).

ELIGIBILITY:
Inclusion Criteria:

* Patient has locally advanced or metastatic stage IIIB/IV Non-small cell lung cancer
* Patient has measurable disease
* Patient has accessible tumor and consents to undergo a tumor biopsy [Part II only]
* Patient is 18 years of age or older
* Patient has a performance status of 0-2 on ECOG scale
* Women of childbearing potential have a negative pregnancy test
* Patients in Part I must: 1. be a female non-smoker with non-squamous histology who has had one or two prior systemic chemotherapies or 2. have documented EGFR mutation or EGFR gene amplification, regardless of demographic or clinical characteristics, who have had no more than two prior systemic chemotherapies.
* Patients in Part II must have had one or two chemotherapy regimens for recurrent or metastatic disease

Exclusion Criteria:

* Patient has had chemotherapy within 2 weeks or biological therapy (e.g. bevacizumab) within 4 weeks
* Patient has not recovered from adverse events from previous therapy within 4 weeks
* Patient has received EGFR-TKI inhibitor/anti-EGFR mAb therapy
* Patient has received IGF1R-TKI inhibitor/anti-IGF1R mAB therapy
* Patient has untreated brain metastases
* Patient has had radiotherapy to a field that affects the chest or abdomen, or thoracic surgery within 3 months prior to entering the study
* Patient is taking part in another clinical study
* Patient abuses drugs or alcohol
* Patient is pregnant or breastfeeding
* Subject is HIV positive
* Patient has active hepatitis
* Patient is using growth hormone or growth hormone inhibitors
* Patient has poorly controlled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Validate imaging platform and molecular markers | FDG response at Weeks 1 and 3 following chemotherapy

SECONDARY OUTCOMES:
Progression-free survival, overall survival | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC